CLINICAL TRIAL: NCT00364663
Title: The Utility and Cost-Effectiveness Analysis of 18-Fluoro-2-Deoxyglucose Positron Emission Tomography in Staging Potential Operable Non-Small Cell Lung Cancer
Brief Title: The Utility and Cost-Effectiveness Analysis of 18F-FDG PETin Staging Potential Operable Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 950307; NSC 95-2314-B-002 -268 -MY2
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2006-08-16 (Estimated); Status verified 2006-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; staging; 18F-FDG PET; decision tree model; cost-effectiveness
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
We plan to conduct a prospective study:

1. to evaluate the accuracy of PET in staging patients with potentially operable non-small cell lung cancer;
2. to evaluate the percentage of futile thoracotomy after PET is introduced in the routine staging modalities for NSCLC patient;
3. to establish a decision tree model based on choices between conventional imaging only and additional PET imaging to analyze their cost-effectiveness.

DETAILED DESCRIPTION:
Lung cancer has been a major health issue worldwide, including Taiwan. According to the data published by the Department of Health, Executive Yuan, Taiwan, 2004, lung cancer is already the leading cause of cancer-related death in Taiwan. Non-small cell lung cancer (NSCLC) represents approximately 75-85% of all primary lung tumors. The strongest prognostic factor for survival is whether the tumor can be completely resected. Surgical resection may be performed for those patients without distant or extended lymph node metastasis. Because of the significant morbidity and mortality for surgical procedure of lung cancer, it is therefore very important to identify and exclude those patients who can't benefit from surgical treatment. Conventional staging, using chest/brain X-ray computed tomography, abdominal echography and radionuclide bone scintigraphy, leads to futile thoracotomies in up to 50% of patients.

Since early 1990s, when 18F-FDG PET has emerged as a promising diagnostic imaging tool in nuclear medicine, a large number of studies have been reported without exception that PET is a better staging tool than CT for patients with NSCLC. However, due to the prohibitive cost, PET is not routinely used for the staging of NSCLC in Taiwan. The extra cost accruing from the introduction of this new technology has been the major concerns from the clinical physicians and health policy makers.

A number of economic evaluation studies overseas have shown that PET is cost-effective in NSCLC when added to conventional work-up. However, due to that the sensitivity and specificity of 18F-FDG PET in staging NSCLC, the cost structure of medical expense, the severity of disease for NSCLC patients when they first present in the hospital, may be different between different countries. To the best of our knowledge, there has been no report that provides a practical guide to introduce PET in staging NSCLC. A cost-effectiveness economic evaluation in Taiwan is thus in demand.

Patient eligibility:

Inclusion criteria: Patients with early NSCLC (stage I & II) Exclusion criteria: (1) patients who are pregnant (2) patients under 18 years old (3) patients who refuse surgical intervention (4) patients who have other known malignancy

ELIGIBILITY:
Inclusion Criteria:

* patients with non-small-cell lung cancer

Exclusion Criteria:

* patients who are pregnant
* patients who are under 18 years old
* patients who do not undergone surgery
* patients who have other known malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Ruoh-Fang Yen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Herder GJ, Verboom P, Smit EF, van Velthoven PC, van den Bergh JH, Colder CD, van Mansom I, van Mourik JC, Postmus PE, Teule GJ, Hoekstra OS. Practice, efficacy and cost of staging suspected non-small cell lung cancer: a retrospective study in two Dutch hospitals. Thorax. 2002 Jan;57(1):11-4. doi: 10.1136/thorax.57.1.11. PMID 11809983
- [Background] Webb WR, Gatsonis C, Zerhouni EA, Heelan RT, Glazer GM, Francis IR, McNeil BJ. CT and MR imaging in staging non-small cell bronchogenic carcinoma: report of the Radiologic Diagnostic Oncology Group. Radiology. 1991 Mar;178(3):705-13. doi: 10.1148/radiology.178.3.1847239.
- [Background] Investigation for mediastinal disease in patients with apparently operable lung cancer. Canadian Lung Oncology Group. Ann Thorac Surg. 1995 Nov;60(5):1382-9. doi: 10.1016/0003-4975(95)00758-d. PMID 8526631
- [Background] van Tinteren H, Hoekstra OS, Smit EF, Verboom P, Boers M; PLUS Study Group. Toward less futile surgery in non-small cell lung cancer? A randomized clinical trial to evaluate the cost-effectiveness of positron emission tomography. Control Clin Trials. 2001 Feb;22(1):89-98. doi: 10.1016/s0197-2456(00)00119-7. PMID 11165427
- [Background] Dwamena BA, Sonnad SS, Angobaldo JO, Wahl RL. Metastases from non-small cell lung cancer: mediastinal staging in the 1990s--meta-analytic comparison of PET and CT. Radiology. 1999 Nov;213(2):530-6. doi: 10.1148/radiology.213.2.r99nv46530. PMID 10551237
- [Background] Yen RF, Chen ML, Liu FY, Ko SC, Chang YL, Chieng PU, Su CT. False-positive 2-[F-18]-fluoro-2-deoxy-D-glucose positron emission tomography studies for evaluation of focal pulmonary abnormalities. J Formos Med Assoc. 1998 Sep;97(9):642-5. PMID 9795534
- [Background] Gambhir SS, Hoh CK, Phelps ME, Madar I, Maddahi J. Decision tree sensitivity analysis for cost-effectiveness of FDG-PET in the staging and management of non-small-cell lung carcinoma. J Nucl Med. 1996 Sep;37(9):1428-36. PMID 8790186